CLINICAL TRIAL: NCT03388294
Title: Evaluation of a Novel Intervention for Infants At Risk for Neurodevelopmental Disorders
Acronym: PIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Southern California (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0292; 1R21HD091547-01 (NIH)
Record Dates: First submitted 2017-12-14; First posted 2018-01-02 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-06

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: communication; sensory; early intervention; parent coaching
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Communication

STUDY DESIGN:
Intervention Model Description: The intervention phases of the study will use a randomized comparative trial design, with two phases. For Study Phase 1, dyads will participate in pretesting; then families will be randomized, stratifying by child age, to one of two treatment arms. Arm 1 families will participate in initial coaching on the PIE sensory reactivity (SR) domain, and Arm 2 families will participate in initial coaching on the PIE prelinguistic communication (PC) domain. Families will participate in 6 weekly coaching sessions in their respective treatment arms, and return for Posttest-1. For Study Phase 2, dyads in Arm 1 will receive 6 weekly coaching sessions on the PC domain, and dyads in Arm 2 will receive 6 weekly coaching sessions on the SR domain. Then families will return for Posttest-2.
Who Masked: Outcomes Assessor
Masking Description: Assessors at all time points after randomization will be blind to the child's treatment arm allocation. Since parents are being coached as part of the intervention, it is not possible to keep them blind to their treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC followed by SR (Experimental): Parents will be coached for 6 weekly sessions in the Parents and Infants Engaged (PIE) intervention pre-linguistic (PC) domain to identify their child's pre-linguistic communication bids during daily routines and respond to those bids in ways that optimize parent-child engagement. After posttest 1, they will be coached for 6 weekly sessions on sensory reactivity bids.
  Interventions: Behavioral: Parents and Infants Engaged
- SR followed by PC (Experimental): Parents will be coached for 6 weekly sessions in the Parents and Infants Engaged (PIE) intervention sensory reactions (SR) domain to identify their child's sensory reactions to daily activities and respond to those reactions or modify the environment in ways that optimize parent-child engagement. After posttest 1, they will be coached for 6 weekly sessions on pre-linguistic communication bids.
  Interventions: Behavioral: Parents and Infants Engaged

INTERVENTIONS:
Behavioral: Parents and Infants Engaged — A novel in-home parent coaching intervention addressing transactions between pre-linguistic communication and sensory reactivity in infants at-risk for autism and other NDs on the one hand, and parent responses to infant cues on the other hand, using live coaching and video feedback methods.
  Other Names: PIE

SUMMARY:
This study entails a "proof of concept" evaluation of a novel intervention, Parents and Infants Engaged (PIE), for prodromal infants at-risk for neurodevelopmental disorders (NDs). The objectives of the current study are to examine whether the PIE intervention (a) transforms parent-infant transactions over time as intended, thereby facilitating increases in the time infants spend in joint engagement with their parents, and (b) is associated with improved social-communication functioning and positive changes in indices of autonomic self-regulation in infants at-risk for NDs.

DETAILED DESCRIPTION:
Rationale:

Providing intervention during infancy, before the full emergence of the symptoms that would lead to a diagnosis of ND based on a behavioral phenotype (e.g., autism spectrum disorder (ASD), language disorder, or attention-deficit/hyperactivity disorder) is supported by 4 premises: (1) The first two years of life are an especially active period of neural development. Due to rapid synaptic proliferation and experientially-influenced shaping of functional connectivity, interventions initiated in infancy may be powerful in promoting more typical neural connectivity (2) Biologically-based differences in infants at-risk for NDs lead to observable differences in sensory reactivity and communication behaviors in most infants by 9-15 months, prior to the full emergence of diagnostic symptoms. (3) Differences in infant behaviors influence the quantity and quality of parent responses. (4) Parent-child transactional processes begin early in infancy and impact long-term child outcomes. Based on these premises, the investigators propose a "proof of concept" evaluation of a novel intervention, Parents and Infants Engaged (PIE), for prodromal infants at-risk for NDs. PIE is designed to directly impact parent responses to behaviors commonly observed in infants at-risk for NDs. Without intervention, these behaviors may fail to elicit parent responses that efficiently scaffold child communication development. Extensive research shows positive associations between caregiver responsiveness and child communication outcomes. Responsiveness is defined by multiple dimensions (i.e., sensitivity, contingency, encouragement, matching interests/activity level, physical affection, quality of language input [e.g., verbal scaffolding], reciprocity, and shared control), which vary within and across caregivers. Children play an active role in eliciting responses from caregivers, emphasizing the co-regulatory or transactional nature of these interactions. This includes biobehavioral co-regulation of arousal levels. Whereas much research comes from studies of typical development, similar transactions occur with young children with NDs. Parent responses vary depending on the preceding behaviors of the child. For example, parents are more likely to respond, and to give a verbal response, to their one-year-olds' gestures than nongestural communicative bids (vocalizations, gaze, actions); also, adults are more likely to respond to infants' speech-like than nonspeech-like vocalizations. Parent responsiveness, in turn, predicts communication outcomes of children with varied NDs.

Aims:

Specific Aim 1: Evaluate the differential changes in attuned parent responsiveness following coaching on two PIE domains - responses to variable infant (a) sensory reactivity (SR) or (b) prelinguistic communication (PC) - as well as cumulative changes in attuned parent responses following coaching on both PIE domains.

Specific Aim 2: Estimate the separate and combined effects of PIE intervention domains on parent-infant engagement and infant-initiated communication with parents.

Specific Aim 3: Determine the extent to which autonomic indices of infant self-regulation change over the course of the PIE intervention.

Recruitment:

To identify infants at-risk for neurodevelopmental disorders, the investigators will use a population-screening method based on birth records in North Carolina, supplemented with distribution of postcards/flyers through physician's offices and public health clinics and email and listserv announcements. Completed First Year Inventories (FYIs) will be scored and screened for risk status. Infants who score at-risk will be flagged, and those families will receive a phone call informing them of the results of the screening (by a qualified/trained project coordinator), and they will be invited for a more comprehensive developmental assessment.

Summary of Measures to be Completed at Each Assessment Time point:

Baseline/Pretest

* Full Mullen Scales of Early Learning (MSEL)
* Sensory Processing Assessment (SPA)
* Brief Observation of Social Communication Change (BOSCC)
* (Respiratory Sinus Arrhythmia (RSA)/ Skin Conductance Level (SCL) Protocol
* Parent-Child Interaction
* Attention Following Protocol
* Sensory Experiences Questionnaire (SEQ)
* MacArthur Bates Communication Development Inventory (MB-CDI)
* Parent Stress Scale

Posttest 1 (6-8 weeks after pretest):

* Parent- Child Interaction
* SEQ

Posttest 2 (13-16 weeks after pretest):

* MSEL Receptive and Expressive Language
* SPA
* BOSCC
* RSA/SCL Protocol
* Parent-Child Interaction
* Attention Following Protocol
* SEQ
* Intervention Rating Profile (intervention group only)

The intervention phases of the study will use a randomized comparative trial design, with two phases. For Intervention Study Phase 1, dyads will participate in the Pretest assessment battery; then the project methodologist will randomize families of eligible infants, stratifying randomization by age (<13 months, 30 days or ≥ 14 months). Families will be randomized to one of two treatment arms: Arm 1 families will participate in initial coaching on the SR domain of PIE, and Arm 2 families will participate in initial coaching on the PC domain of PIE. Families will participate in 6 coaching sessions in their respective treatment arms, and then return for Posttest-1 (to test the separate impacts of the PIE content domains on parent responses and infant outcomes). For Intervention Study Phase 2, dyads in Arm 1, will receive 6 coaching sessions on the PC domain, and dyads in Arm 2 will receive 6 coaching sessions on the SR domain; coaching for each group will also review their respective content domain coached in Intervention Study Phase 1. Then families will return for Posttest-2 (to evaluate the effects of the full PIE intervention).

Due to COVID-19 restrictions, intervention may be carried out via video-conference platform for no more than one session. Parent-report questionnaires only will be collected in lieu of in-person assessments for Posttest-2 for participants unable to attend in-person.

Data Analyses:

All data will be cleaned and inspected for outliers, missing data and distributional irregularities. Where error distributions potentially deviate from normality, or heteroscedasticity is suspected, the tests of the contrasts will be conducted using exact (resampling-based) nonparametric methods. Proportional outcomes will be arc sin transformed before entering them into the models. For the frequency count outcome, if counts are not sufficiently large (e.g., ≥ 8) that a normal approximation to a Poisson error distribution is appropriate, Poisson or negative binomial regression methods or nonparametric approaches may be employed.

All primary analyses will be conducted to explore a priori contrasts of interest within a repeated measures framework. Of primary interest will be the contrast of Pretest to Posttest-1 scores and the contrast of Pretest to Posttest-2 scores (time effect). In addition, the models will include terms for treatment arm effects and treatment arm-by-time interactions.

At Posttest-1, the investigators anticipate statistically significant time, treatment arm, and arm-by-time interactions, with parents showing differentially greater attuned responses to infant SR or PC, consistent with their respective treatment arm. By Posttest-2, however, the investigators predict group equivalence in responsiveness, with no differential time effects. A follow-up test of the contrast between Posttest-1 and Posttest-2 will verify that parents in Arm 1 maintained their attuned SR responsiveness gains, while parents in Arm 2 "caught up" on attuned SR responsiveness, and vice versa for PC attunement. For H2a, the investigators expect increases in joint engagement from Pretest to Posttest-1, with additional increases at Posttest-2 (time effects), and no differential treatment arm effects or interactions at either Posttest. For H2b, the investigators anticipate minimal increases in infant intentional communication at Posttest-1 in either treatment arm, with comparable improvements (time effects) in each group at Posttest-2. Similarly, on the physiological measures addressing H3a (measured only at Pretest and Posttest-2) the investigators anticipate comparable improvements in RSA and SCL (time effect) in both arms.

Although the investigators are performing multiple statistical tests across outcomes and hypotheses in addressing the specific aims, in this project it is more important to avoid overlooking statistical signals of effectiveness of the innovative PIE intervention approach (Type II errors), than avoiding false assertions of effectiveness (Type I errors). The investigators believe it is premature, therefore, to employ conservative adjustments to the Type I error rates in statistical tests, which would compromise the power of statistical tests to detect such signals. Assuming recruitment of 44 infant-parent dyads and allowing for a 9% (n=4) dropout rate, which is consistent with high retention rates (> 95%) in our prior intervention studies, 40 dyads (20 per treatment arm) will have complete data for analyses. Assuming a conventional Type I error rate of .05, and intercorrelations among the repeated measures from .3 to .7, the magnitude of treatment group effects detectable with a .80 statistical power will range from f=.37 to .42, respectively, which are large standardized effects. The magnitude of time effects and time-by-treatment arm interaction effects detectable with a .80 power will range from .27 to .18, also respectively, which are medium-sized standardized effects. Thus, the study is underpowered to detect any but large differences between the treatment arms and medium-sized or larger effects on time and time-by treatment arm interactions. More importantly than the statistical comparisons, though, the analyses will yield key descriptive characterizations of the treatment-arm effects at the two posttest points (i.e.,means, medians, proportions, and variances) on key outcomes, as well as effect size estimates that can be used in planning a larger scaled efficacy trial of the PIE intervention.

ELIGIBILITY:
Inclusion Criteria:

* For the intervention trial: infant must meet risk criteria on the First Years Inventory (Calculated based on data collected in another study where risk status on the FYI was confirmed with follow up at 3 years. We empirically determined combinations of the two FYI domain scores that would sort respondents into "at-risk" and "not-at-risk." The resulting cut-points enabled us to sort children such that we capture about 1/3 of those who would go on to be confirmed as having a autism spectrum diagnosis while misclassifying less than 5% of the typically developing (TD) sample as at-risk). Infants also must score at least one s.d. below the mean on either the Receptive or Expressive subscale t scores AND meet the following SPA inclusion criteria on hyporeactivity (HYPO) or hyperreactivity (HYPER):

  * "HYPO": Cut-point (equal or greater than) of 1.69 for Mean of the raw orienting score across 7 items, each with the range of 1 to 4 possible points)
  * "HYPER": Cut-point (equal or greater than) of .333 for Mean of the raw approach/avoid novel toys score across 9 items, each with the range of 0 to 2 possible points) OR Any clear "defensive" response on orienting items or "Yes" to covering ears to sound (in stereotypies checklist)

Exclusion Criteria:

* families who speak English < 50% of the time at home
* infants with previously identified genetic disorders (e.g., Down syndrome)
* infants with identified vision/hearing/physical impairments.

Ages: 11 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace T Baranek, PhD, Principal Investigator — University of Southern California; Linda R Watson, EdD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tamis-LeMonda CS, Kuchirko Y, Song L. Why is infant language learning facilitated by parental responsiveness? Current Directions in Psychological Science. 2014;23(2):121-126.
- [Background] Baranek GT, Watson LR, Turner-Brown L, Field SH, Crais ER, Wakeford L, Little LM, Reznick JS. Preliminary efficacy of adapted responsive teaching for infants at risk of autism spectrum disorder in a community sample. Autism Res Treat. 2015;2015:386951. doi: 10.1155/2015/386951. Epub 2015 Jan 11. PMID 25648749
- [Background] Watson LR, Baranek GT, Roberts JE, David FJ, Perryman TY. Behavioral and physiological responses to child-directed speech as predictors of communication outcomes in children with autism spectrum disorders. J Speech Lang Hear Res. 2010 Aug;53(4):1052-64. doi: 10.1044/1092-4388(2009/09-0096). Epub 2010 Jul 14. PMID 20631229
- [Background] Turner-Brown LM, Baranek GT, Reznick JS, Watson LR, Crais ER. The First Year Inventory: a longitudinal follow-up of 12-month-old to 3-year-old children. Autism. 2013 Sep;17(5):527-40. doi: 10.1177/1362361312439633. Epub 2012 Jul 10. PMID 22781058
- [Background] Guthrie W, Swineford LB, Nottke C, Wetherby AM. Early diagnosis of autism spectrum disorder: stability and change in clinical diagnosis and symptom presentation. J Child Psychol Psychiatry. 2013 May;54(5):582-90. doi: 10.1111/jcpp.12008. PMID 23078094
- [Background] Barnett MA, Gustafsson H, Deng M, Mills-Koonce WR, Cox M. Bidirectional Associations Among Sensitive Parenting, Language Development, and Social Competence. Infant Child Dev. 2012 Jul;21(4):374-393. doi: 10.1002/icd.1750. PMID 25126021
- [Background] Mahoney G, Perales F. Relationship-focused early intervention with children with pervasive developmental disorders and other disabilities: a comparative study. J Dev Behav Pediatr. 2005 Apr;26(2):77-85. doi: 10.1097/00004703-200504000-00002. PMID 15827458
- [Background] Kochanska G, Forman DR, Aksan N, Dunbar SB. Pathways to conscience: early mother-child mutually responsive orientation and children's moral emotion, conduct, and cognition. J Child Psychol Psychiatry. 2005 Jan;46(1):19-34. doi: 10.1111/j.1469-7610.2004.00348.x. PMID 15660641
- [Background] Sameroff AJ, Mackenzie MJ. Research strategies for capturing transactional models of development: the limits of the possible. Dev Psychopathol. 2003 Summer;15(3):613-40. doi: 10.1017/s0954579403000312. PMID 14582934
- [Background] Baker JK, Fenning RM, Howland MA, Baucom BR, Moffitt J, Erath SA. Brief Report: A Pilot Study of Parent-Child Biobehavioral Synchrony in Autism Spectrum Disorder. J Autism Dev Disord. 2015 Dec;45(12):4140-6. doi: 10.1007/s10803-015-2528-0. PMID 26183724
- [Background] Feldman R. Mutual influences between child emotion regulation and parent-child reciprocity support development across the first 10 years of life: Implications for developmental psychopathology. Dev Psychopathol. 2015 Nov;27(4 Pt 1):1007-23. doi: 10.1017/S0954579415000656. PMID 26439059
- [Background] Hill-Soderlund AL, Mills-Koonce WR, Propper C, Calkins SD, Granger DA, Moore GA, Gariepy JL, Cox MJ. Parasympathetic and sympathetic responses to the strange situation in infants and mothers from avoidant and securely attached dyads. Dev Psychobiol. 2008 May;50(4):361-76. doi: 10.1002/dev.20302. PMID 18393278
- [Background] Baranek GT. Autism during infancy: a retrospective video analysis of sensory-motor and social behaviors at 9-12 months of age. J Autism Dev Disord. 1999 Jun;29(3):213-24. doi: 10.1023/a:1023080005650. PMID 10425584
- [Background] Ben-Sasson A, Carter AS. The contribution of sensory-regulatory markers to the accuracy of ASD screening at 12 months. Research in Autism Spectrum Disorders. 2013;7(7):879-888.
- [Background] Watson LR, Crais ER, Baranek GT, Dykstra JR, Wilson KP. Communicative gesture use in infants with and without autism: a retrospective home video study. Am J Speech Lang Pathol. 2013 Feb;22(1):25-39. doi: 10.1044/1058-0360(2012/11-0145). Epub 2012 Jul 30. PMID 22846878
- [Background] Beauchaine TP, Gatzke-Kopp L, Neuhaus E, Chipman J, Reid MJ, Webster-Stratton C. Sympathetic- and parasympathetic-linked cardiac function and prediction of externalizing behavior, emotion regulation, and prosocial behavior among preschoolers treated for ADHD. J Consult Clin Psychol. 2013 Jun;81(3):481-493. doi: 10.1037/a0032302. Epub 2013 Apr 1. PMID 23544677
- [Background] Lam-Cassettari C, Wadnerkar-Kamble MB, James DM. Enhancing Parent-Child Communication and Parental Self-Esteem With a Video-Feedback Intervention: Outcomes With Prelingual Deaf and Hard-of-Hearing Children. J Deaf Stud Deaf Educ. 2015 Jul;20(3):266-74. doi: 10.1093/deafed/env008. Epub 2015 Mar 28. PMID 25819293
- [Background] Hoivik MS, Lydersen S, Drugli MB, Onsoien R, Hansen MB, Nielsen TS. Video feedback compared to treatment as usual in families with parent-child interactions problems: a randomized controlled trial. Child Adolesc Psychiatry Ment Health. 2015 Feb 12;9:3. doi: 10.1186/s13034-015-0036-9. eCollection 2015. PMID 25699090
- [Background] Beauchaine TP, Neuhaus E, Gatzke-Kopp LM, Reid MJ, Chipman J, Brekke A, Olliges A, Shoemaker S, Webster-Stratton C. Electrodermal responding predicts responses to, and may be altered by, preschool intervention for ADHD. J Consult Clin Psychol. 2015 Apr;83(2):293-303. doi: 10.1037/a0038405. Epub 2014 Dec 8. PMID 25486374
- [Background] Baranek GT, Watson LR, Crais E, Reznick S. First-year inventory (FYI) 2.0. University of North Carolina at Chapel Hill; 2003.
- [Background] Watson LR, Patten E, Baranek GT, Poe M, Boyd BA, Freuler A, Lorenzi J. Differential associations between sensory response patterns and language, social, and communication measures in children with autism or other developmental disabilities. J Speech Lang Hear Res. 2011 Dec;54(6):1562-76. doi: 10.1044/1092-4388(2011/10-0029). Epub 2011 Aug 23. PMID 21862675
- [Background] Watson LR, Roberts JE, Baranek GT, Yoder P. Respiratory sinus arrhythmia as a predictor of language outcomes in children with autism. International Journal of Psychophysiology. 2012;85(3):348. Accessed 9/28/2015 2:41:37 PM.
- [Background] Grzadzinski R, Carr T, Colombi C, McGuire K, Dufek S, Pickles A, Lord C. Measuring Changes in Social Communication Behaviors: Preliminary Development of the Brief Observation of Social Communication Change (BOSCC). J Autism Dev Disord. 2016 Jul;46(7):2464-79. doi: 10.1007/s10803-016-2782-9. PMID 27062034

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Dyads
Groups:
- PC Followed by SR: Parents will first be coached to respond to their infant's pre-linguistic communication (PC) cues. After posttest 1, they will be coached in responding to the infant's sensory reactivity (SR) cues.
  Parents and Infants Engaged (PIE): A parent coaching intervention addressing transactions between pre-linguistic communication and sensory reactivity in infants at-risk for autism and other neurodevelopmental disorders (NDs) on the one hand, and parent responses to infant cues on the other hand.
- SR Followed by PC: Parents will first be coached to respond to their infant's sensory reactivity (SR) cues. After posttest 1, they will be coached in responding to the infant's pre-linguistic communication (PC) cues.
  Parents and Infants Engaged (PIE): A parent coaching intervention addressing transactions between pre-linguistic communication and sensory reactivity in infants at-risk for autism and other neurodevelopmental disorders (NDs) on the one hand, and parent responses to infant cues on the other hand.
Period: Overall Study
Arm/Group | PC Followed by SR | SR Followed by PC
Started | 42; 21 Dyads | 30; 15 Dyads
Posttest 1 | 38; 19 Dyads | 30; 15 Dyads
Posttest 2 | 38; 19 Dyads | 30; 15 Dyads
Completed | 38; 19 Dyads | 30; 15 Dyads
Not Completed | 4; 2 Dyads | 0; 0 Dyads

BASELINE CHARACTERISTICS:
Units Other Than Participants: Dyads
Groups:
- PC Followed by SR: Using the PIE intervention, parents will first be coached to respond to their infant's pre-linguistic communication cues. After posttest 1, they will be coached in responding to the infant's sensory reactivity cues.
- SR Followed by PC: Using the PIE intervention, parents will first be coached to respond to their infant's sensory reactivity cues. After posttest 1, they will be coached in responding to the infant's pre-linguistic communication cues.
- Total: Total of all reporting groups
Arm/Group | PC Followed by SR | SR Followed by PC | Total
Number analyzed (Participants) | 42 | 30 | 72
Number analyzed (Dyads) | 21 | 15 | 36
Age, Customized [Mean (Standard Deviation); unit: Months] — Infant age at Baseline assessment adjusted for prematurity for those born =/< 36 weeks gestational age. Population: Parent age data unavailable.
  Months
    number analyzed (Participants) | 21 | 15 | 36
    Infant age | 13.95 (1.66) | 14.07 (1.67) | 14.00 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender reported separately for parent/caregiver and infants.
  Participants
    number analyzed (Participants) | 21 | 15 | 36
    Infants: Female | 7 | 3 | 10
    Infants: Male | 14 | 12 | 26
    Parents/Caregivers: Female | 17 | 14 | 31
    Parents/Caregivers: Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data reported separately for parent/caregiver and infants.
  Participants
    number analyzed (Participants) | 21 | 15 | 36
    Infants: Hispanic or Latino | 5 | 2 | 7
    Infants: Not Hispanic or Latino | 15 | 13 | 28
    Infants: Unknown or Not Reported | 1 | 0 | 1
    Parents/Caregivers: Hispanic or Latino | 3 | 3 | 6
    Parents/Caregivers: Not Hispanic or Latino | 14 | 10 | 24
    Parents/Caregivers: Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race reported separately for parent/caregiver and infants.
  Participants
    number analyzed (Participants) | 21 | 15 | 36
    Infants: American Indian or Alaska Native | 0 | 0 | 0
    Infants: Asian | 1 | 1 | 2
    Infants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Infants: Black or African American | 2 | 2 | 4
    Infants: White | 13 | 12 | 25
    Infants: More than one race | 3 | 0 | 3
    Infants: Unknown or Not Reported | 2 | 0 | 2
    Parents/Caregivers: American Indian or Alaska Native | 1 | 0 | 1
    Parents/Caregivers: Asian | 1 | 0 | 1
    Parents/Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parents/Caregivers: Black or African American | 1 | 1 | 2
    Parents/Caregivers: White | 12 | 11 | 23
    Parents/Caregivers: More than one race | 2 | 0 | 2
    Parents/Caregivers: Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 30 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Percent of Parent Child Dyadic Engagement Over Time From Baseline to Posttest 1
Description: This system entails continuous coding of infants' attention engagement into one of 6 mutually exclusive states: unengaged, onlooking, object engaged, person-engaged, supported joint engagement, and coordinated joint engagement. Due to the importance of the construct of engagement to our PIE theory of change, the total percent of time in dyadic engagement (higher level supported + coordinated) will serve as the most proximal intervention outcome (i.e., changes expected at Posttest-1). Recent studies with children with NDs have shown that the coding system is sensitive to change in joint engagement after relatively short interventions.
Time Frame: Baseline, Posttest 1 (6-8 weeks after baseline)
Population: Four dyads in the PC followed by SR and 1 dyad in the SR followed by PC were unavailable at Posttest 1
Measure: Mean (Standard Deviation); unit: percent time in dyadic engagement
Units Other Than Participants: Dyads
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 42 | 30
Number analyzed (Dyads) | 21 | 15
percent time in dyadic engagement
  Baseline | 22.01 (13.63) | 16.91 (9.70)
  Posttest 1: number analyzed (Participants) | 34 | 28
  Posttest 1: number analyzed (Dyads) | 17 | 14
  Posttest 1 | 26.55 (14.62) | 27.09 (7.81)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.028, Mixed Models Analysis; Mean Difference (Net) = 7.32

2. Primary Outcome: Change in Mean Percent of Parent Child Dyadic Engagement Over Time From Baseline to Posttest 2
Description: as for outcome 1
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Three dyads in the PC followed by SR and 2 dyads in the SR followed by PC were unavailable at Posttest 2
Measure: Mean (Standard Deviation); unit: percent time in dyadic engagement
Units Other Than Participants: Dyads
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 42 | 30
Number analyzed (Dyads) | 21 | 15
percent time in dyadic engagement
  Baseline | 22.01 (13.63) | 16.91 (9.70)
  Posttest 2: number analyzed (Participants) | 36 | 26
  Posttest 2: number analyzed (Dyads) | 18 | 13
  Posttest 2 | 30.12 (16.78) | 35.23 (22.12)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; The focus for this analysis is change over time; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 12.75

3. Secondary Outcome: Change in Rating of Parent Responsiveness to Child Sensory Reactivity Cues From Baseline to Posttest 1
Description: Parent-child interaction videos will be coded for parent responsiveness to child sensory reactivity cues. These are each rated on a 0-7 scale. Higher scores indicate greater responsivity from parents.
Time Frame: Baseline, Posttest 1 (6-8 weeks after baseline)
Population: Data for 1 enrolled parent was unavailable at Baseline and data 3 enrolled parents were unavailable at Posttest 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 20 | 15
score on a scale
  Baseline | 3.73 (1.15) | 3.47 (0.76)
  Posttest 1: number analyzed (Participants) | 18 | 15
  Posttest 1 | 4.33 (0.98) | 4.02 (1.35)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Superiority; p = 0.87, Mixed Models Analysis

4. Secondary Outcome: Change in Rating of Parent Responsiveness to Child Sensory Reactivity Cues From Baseline to Posttest 2
Description: as for outcome 3
Time Frame: Baseline, posttest 2 (13-16 weeks after baseline)
Population: Data for 1 enrolled parent was unavailable at Baseline and data 3 enrolled parents were unavailable at Posttest 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 20 | 15
score on a scale
  Baseline | 3.73 (1.15) | 3.47 (0.76)
  Posttest 2: number analyzed (Participants) | 19 | 14
  Posttest 2 | 4.03 (0.93) | 4.39 (1.21)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.006, Mixed Models Analysis; Mean Difference (Net) = 0.61

5. Secondary Outcome: Change in Rating of Parent Responsiveness to Child Prelinguistic Communication Cues From Baseline to Posttest 1
Description: Parent-child interaction videos will be coded for parent responsiveness to child prelinguistic communication cues. These are each rated on a 0-7 scale. Higher scores indicate greater responsivity from parents.
Time Frame: Baseline, Posttest 1 (6-8 weeks after pretest)
Population: Data for 4 enrolled parents was unavailable at Posttest 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline | 4.04 (0.90) | 4.57 (1.23)
  Posttest 1: number analyzed (Participants) | 17 | 15
  Posttest 1 | 4.54 (0.97) | 4.88 (0.92)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Superiority; p = 0.76, Mixed Models Analysis

6. Secondary Outcome: Change in Rating of Parent Responsiveness to Child Prelinguistic Communication Cues From Baseline to Posttest 2
Description: as for outcome 5
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Data for 4 enrolled parents was unavailable at Posttest 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline | 4.04 (0.90) | 4.57 (1.23)
  Posttest 2: number analyzed (Participants) | 18 | 14
  Posttest 2 | 4.39 (1.06) | 4.32 (0.95)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.849, Mixed Models Analysis

7. Secondary Outcome: Change in Rate of Infant Intentional Communication Over Time, Baseline to Posttest 1
Description: Rate of child intentional communication during parent-child interaction, coded from videos. Video recordings of parent-child interactions were coded for infants' intentional communication acts (i.e., acts directed to the parent): vocalizations, gestures, or both (acts combining vocalizations and gestures). A total acts variable was calculated for the sum of all communication acts in a recording. The total communication acts variable was transformed into a rate variable (instances per minute) for the purpose of this outcome.
Time Frame: Baseline, Posttest 1 (6-8 weeks after pretest)
Population: Data for 3 enrolled children was unavailable at Posttest 1
Measure: Mean (Standard Deviation); unit: instances per minute
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
instances per minute
  Baseline | 0.48 (0.44) | 0.48 (0.38)
  Posttest 1: number analyzed (Participants) | 18 | 15
  Posttest 1 | 0.71 (0.64) | 0.67 (0.66)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.063, Mixed Models Analysis; Mean Difference (Net) = 0.20

8. Secondary Outcome: Change in Rate of Infant Intentional Communication Over Time, Baseline to Posttest 2
Description: Rate of infant intentional communication during parent-child interaction, coded from videos. Video recordings of parent-child interactions were coded for infants' intentional communication acts (i.e., acts directed to the parent): vocalizations, gestures, or both (acts combining vocalizations and gestures). A total acts variable was calculated for the sum of all communication acts in a recording. The total communication acts variable was transformed into a rate variable (instances per minute) for the purpose of this outcome.
Time Frame: Baseline, Posttest 2 (13-16 weeks after pretest)
Population: Data for 4 enrolled children were unavailable for Posttest 2
Measure: Mean (Standard Deviation); unit: instances per minute
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
instances per minute
  Baseline | 0.48 (0.44) | 0.48 (0.38)
  Posttest 2: number analyzed (Participants) | 18 | 14
  Posttest 2 | 0.92 (0.53) | 1.03 (0.70)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.48

9. Secondary Outcome: Change in Respiratory Sinus Arrhythmia From Baseline to Posttest 2 During Social Stimuli
Description: Respiratory Sinus Arrhythmia (RSA) levels will be collected using a standard protocol while the child is seated in a high chair exposed to social and non-social stimuli. RSA indexes the variability in heartrate that is associated with respiratory inspiration and expiration. RSA levels are expected to increase with development during exposure to both social and nonsocial stimuli in the context of this protocol. Higher RSA levels during exposure to social stimuli involving child-directed speech have been predictive of better language outcomes in previous studies of preschoolers diagnosed with autism.
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Due to challenges getting infants to keep electrodes attached or remain still during procedure, some did not have data available for Baseline but did have data for Posttest 2 and vice versa. Data were unavailable for 15 enrolled children at Baseline and 21 enrolled children for Posttest 2.
Measure: Mean (Standard Deviation); unit: ln(ms^2)
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 19 | 10
ln(ms^2)
  Baseline: number analyzed (Participants) | 14 | 7
  Baseline | 4.07 (1.07) | 4.54 (0.94)
  Posttest 2: number analyzed (Participants) | 10 | 5
  Posttest 2 | 4.52 (1.19) | 4.25 (1.07)

10. Secondary Outcome: Change in Respiratory Sinus Arrhythmia From Baseline to Posttest 2 During Non-Social Stimuli
Description: as for outcome 9
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Due to challenges getting infants to keep electrodes attached or remain still during procedure, some did not have data available for Baseline but did have data for Posttest 2 and vice versa. Data were unavailable for 15 enrolled children at Baseline and 20 enrolled children for Posttest 2.
Measure: Mean (Standard Deviation); unit: ln(ms^2)
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 19 | 10
ln(ms^2)
  Baseline: number analyzed (Participants) | 14 | 7
  Baseline | 3.81 (0.96) | 4.24 (1.10)
  Posttest 2: number analyzed (Participants) | 10 | 6
  Posttest 2 | 4.36 (1.35) | 3.61 (4.24)

11. Secondary Outcome: Change in Skin Conductance Levels From Baseline to Posttest 2
Description: Skin conductance levels will be collected using a standard protocol while the child is seated in a high chair exposed to social and non-social stimuli.
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Excessive movement artifacts in skin conductance data prevented derivation of valid skin conductance levels from children
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in The Behavioral Observation of Social Communication Change (BOSCC) From Baseline to Posttest 2
Description: A treatment response measure of social communication behaviors and other behaviors associated with autism spectrum disorder (ASD). Administration of the BOSCC involves a 12-minute video recorded interaction between an examiner and a young child using two standard sets of toys and play with bubbles. Behaviors are coded from video. Total score range is 16-80. Higher scores indicate more atypical social communication skills, lower scores indicate better skills.
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Some video durations were too short to qualify for scoring per BOSCC protocol. Data were unavailable for 7 enrolled children at Baseline and 8 enrolled children for Posttest 2. The majority of enrolled children (i.e., 25) had data available at both timepoints; 4 enrolled children had data at Baseline only; 3 enrolled children at Posttest 2 only; and 4 enrolled children had no data available at either timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 18 | 14
score on a scale
  Baseline: number analyzed (Participants) | 16 | 13
  Baseline | 34.06 (4.17) | 30.96 (5.22)
  Posttest 2: number analyzed (Participants) | 15 | 13
  Posttest 2 | 29.40 (6.47) | 29.62 (6.83)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.036, Mixed Models Analysis; Mean Difference (Net) = -2.90

13. Secondary Outcome: Change in The Attention Following Protocol (AF Protocol) From Baseline to Posttest 2
Description: Designed to measure the extent to which children will follow attentional cues of the examiner. Six prompts for attention following are embedded into the larger study protocol. Items are scored dichotomously as yes "1" or no "0".Total score range is 0-6. Higher scores indicate more typical responses to bids for joint attention.
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Data were unavailable for enrolled child at Baseline and 4 enrolled children at Posttest 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 14
score on a scale
  Baseline | 2.14 (2.08) | 2.93 (2.37)
  Posttest 2: number analyzed (Participants) | 18 | 14
  Posttest 2 | 3.78 (2.34) | 4.00 (2.25)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.0002, Mixed Models Analysis

14. Secondary Outcome: Change in Mullen Scales of Early Learning Receptive Language T-Scores From Baseline to Posttest 2
Description: The Mullen Scales of Early Learning (MSEL) is a standardized developmental assessment for children birth to 58 months, frequently used in studies of children with NDs, This outcome comprises changes in standardized T-scores (Mean = 50, SD = 10) on the MSEL Receptive Language scale. Higher scores indicate greater developmental skills.
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Data were unavailable for 4 enrolled children at Posttest 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline | 30.19 (8.73) | 34.33 (12.72)
  Posttest 2: number analyzed (Participants) | 18 | 14
  Posttest 2 | 30.56 (10.89) | 33.71 (13.79)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.864, Mixed Models Analysis; Mean Difference (Net) = 0.36

15. Secondary Outcome: Change in Mullen Scales of Early Learning Expressive Language T-scores From Baseline to Posttest 2
Description: The MSEL is a standardized developmental assessment for children birth to 58 months, frequently used in studies of children with NDs, This outcome comprises changes in standardized T-scores (Mean = 50, SD = 10) on the MSEL Expressive Language scale. Higher scores indicate greater developmental skills.
Time Frame: Baseline, posttest 2 (13-16 weeks after baseline)
Population: Data were unavailable for 4 enrolled children at Posttest 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline | 32.38 (8.84) | 32.93 (11.11)
  Posttest 2: number analyzed (Participants) | 18 | 14
  Posttest 2 | 34.06 (9.36) | 37.29 (11.92)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.12, Mixed Models Analysis; Mean Difference (Net) = 3.14

16. Secondary Outcome: Change in Sensory Processing Assessment for Young Children From Baseline to Posttest 2 in Hypo-Reactivity
Description: A play-based assessment used to measure children's approach-avoidance to novel sensory toys (i.e., hyper-reactivity) and orienting responses (i.e., hypo-reactivity) across three sensory modalities (auditory, visual, tactile). The investigators will report a mean score for Hypo (range = 1-5) and Hyper (range = 1-5) sensory subscales. Higher scores indicate greater sensory differences in that domain (e.g. a high hypo domain score would indicate more hyposensitive reactions to sensory stimuli seen in the child).
Time Frame: Baseline, posttest 2 (13-16 weeks after baseline)
Population: Data were unavailable for 4 enrolled children at Baseline and 6 enrolled children at Posttest 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline: number analyzed (Participants) | 19 | 13
  Baseline | 2.58 (0.68) | 2.10 (0.85)
  Posttest 2: number analyzed (Participants) | 17 | 13
  Posttest 2 | 2.61 (0.91) | 1.99 (0.72)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.881, Mixed Models Analysis; Mean Difference (Net) = 0.02

17. Secondary Outcome: Change in Sensory Processing Assessment for Young Children From Baseline to Posttest 2 in Hyper-Reactivity
Description: as for outcome 16
Time Frame: Baseline, posttest 2 (13-16 weeks after baseline)
Population: Data were unavailable for 4 enrolled children at Baseline and 6 enrolled children at Posttest 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline: number analyzed (Participants) | 19 | 13
  Baseline | 1.66 (0.39) | 1.55 (0.40)
  Posttest 2: number analyzed (Participants) | 17 | 13
  Posttest 2 | 1.59 (0.33) | 1.59 (0.35)
Statistical Analysis 1: Comparison: PC Followed by SR vs SR Followed by PC; Test type: Other — The focus for this analysis is change over time; p = 0.846, Mixed Models Analysis; Mean Difference (Net) = 0.02

18. Secondary Outcome: Change in The Sensory Experiences Questionnaire Version 2.1 From Baseline to Posttest 1 in Hypo-reactivity
Description: A 43 item parent questionnaire that asks about the child's responses to various sensory stimuli in the context of functional activities and daily routines in the child's environment. It also documents strategies parents use to respond to their child's behaviors. Hyper and Hypo mean domain scores will be reported (range = 1-5). Greater domain scores indicate a greater presence of that type of sensory response.
Time Frame: Baseline, posttest 1 (6-8 weeks after baseline)
Population: No data are available for 3 enrolled children at Baseline and 16 at Posttest 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline: number analyzed (Participants) | 19 | 14
  Baseline | 2.18 (0.62) | 1.92 (0.69)
  Posttest 1: number analyzed (Participants) | 11 | 9
  Posttest 1 | 2.26 (0.57) | 2.04 (0.74)

19. Secondary Outcome: Change in The Sensory Experiences Questionnaire Version 2.1 From Baseline to Posttest 1 in Hyper-reactivity
Description: as for outcome 18
Time Frame: Baseline, posttest 1 (6-8 weeks after baseline)
Population: Data were unavailable for 3 enrolled children at Baseline and 16 at Posttest 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline: number analyzed (Participants) | 19 | 14
  Baseline | 2.03 (0.34) | 1.81 (0.33)
  Posttest 1: number analyzed (Participants) | 11 | 9
  Posttest 1 | 1.92 (0.39) | 1.85 (0.29)

20. Secondary Outcome: Change in The Sensory Experiences Questionnaire Version 2.1 From Baseline to Posttest 2 in Hypo-reactivity
Description: as for outcome 18
Time Frame: Baseline, posttest 2 (13-16 weeks after baseline)
Population: Data were unavailable for 3 enrolled participants at Baseline and 16 at Posttest 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline: number analyzed (Participants) | 19 | 14
  Baseline | 2.18 (0.62) | 1.92 (0.69)
  Posttest 2: number analyzed (Participants) | 12 | 8
  Posttest 2 | 2.31 (0.85) | 2.27 (0.70)

21. Secondary Outcome: Change in The Sensory Experiences Questionnaire Version 2.1 From Baseline to Posttest 2 in Hyper-reactivity
Description: as for outcome 18
Time Frame: Baseline, Posttest 2 (13-16 weeks after baseline)
Population: Data are unavailable for 3 enrolled children at Baseline and 16 at Posttest 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC Followed by SR | SR Followed by PC
Number analyzed (Participants) | 21 | 15
score on a scale
  Baseline: number analyzed (Participants) | 19 | 14
  Baseline | 2.03 (0.34) | 1.81 (0.33)
  Posttest 2: number analyzed (Participants) | 12 | 8
  Posttest 2 | 1.92 (0.22) | 2.21 (0.59)

ADVERSE EVENTS:
Time Frame: From signing Informed Consent through Posttest 2, a total of approximately 4 months.
Arm/Group | PC Followed by SR | SR Followed by PC
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/30
Other Adverse Events (participants affected / at risk) | 0/42 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03388294/Prot_SAP_000.pdf